CLINICAL TRIAL: NCT02189161
Title: A Safety and Tolerability Trial of Circumferential Anal Canal Radiofrequency Ablation For Anal Intraepithelial Neoplasia Using the Barrx™ Ablation System
Brief Title: A Safety and Tolerability of Circumferential Anal Canal Radiofrequency Ablation For Anal Intraepithelial Neoplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-253
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Anal Intraepithelial Neoplasia (AIN); High-grade Squamous Intraepithelial Lesions (HSIL)
Keywords: anal intraepithelial neoplasia; AIN; Radiofrequency Ablation; RFA
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiofrequency Ablation (Experimental): circumferential radiofrequency ablation (RFA) to the anal canal
  Interventions: Device: Radiofrequency Ablation (Barrx™)

INTERVENTIONS:
Device: Radiofrequency Ablation (Barrx™) — Anal canal RFA is performed to the full anal canal, 3 cm above the dentate line to the anocutaneous line proximal to the verge. The procedure entails Barrx60 ablation device, introducing the device into the anus through the anoscope, placing the electrode surface in contact with the target tissue and delivering 3 bursts of energy in rapid succession at an energy density setting of 12 J/cm2.
  Other Names: Barrx™ Ablation System

SUMMARY:
Assess the safety, feasibility, and patient tolerability of circumferential radiofrequency ablation (RFA) to the anal canal for patients with anal intraepithelial neoplasia (AIN). Patients will have AIN with high grade squamous intraepithelial lesions (HSIL) and the RFA will be applied using the Barrx™ Ablation System.

ELIGIBILITY:
Inclusion Criteria

Candidates for this study must meet all of the following criteria:

1. Age 18-75 years
2. HRA 2 to 8 weeks prior to the 0 month RFA visit yielding one or more flat, non-condylomatous biopsy-proven HSILs that are

   * Located entirely within the eligible treatment zone AND
   * Contiguous with the squamocolumnar junction
3. Eligible treatment zone (ETZ) is defined as

   * 3 cm above the dentate line to the anocutaneous line AND
   * Full anorectal circumference
4. If female of child-bearing age, negative pregnancy test within 8 weeks of the 0 month RFA visit and declared intent to remain on birth control throughout the trial, or declaration of infertility defined as subject report of status as post-menopausal or surgically sterile (status post hysterectomy or tubal ligation).
5. If HIV positive

   * HIV positive on antiretroviral therapy for at least 3 months with laboratory blood work within 12 weeks prior to the 0 month visit demonstrating viral load < 50
   * CD4 count ≥ 250/mm3
   * ANC > 750/mm3
   * Platelet count ≥ 75,000/mm3
   * Hemoglobin ≥ 9.0 g/dl
   * INR and PTT normal

Exclusion Criteria

Candidates will be ineligible for enrollment in the study if any of the following conditions apply:

1. Any biopsy-proven HSIL partially outside of the ETZ (for example, an HSIL lesion with extension to the perianal skin)
2. Any condylomas in the eligible treatment zone > 1/2 cm diameter

   • Note: Condylomas in the eligible treatment zone < 1/2 cm in diameter must be excised or cauterized (not treated topically) before or during Visit 1 (0 month RFA visit)
3. Any anal or rectal pathology requiring treatment including ulcer, fistula, fissure, or proctitis
4. Any anal stricture or stenosis in patient history or upon examination.
5. Symptomatic scarring in anal canal (i.e. not pliable, hyperkeratosis)
6. History of or present anal or rectal cancer
7. History of pelvic radiation therapy
8. History of HPV vaccination or plans to initiate HPV vaccination during the trial
9. History of ablation or resection therapy within the ETZ within 6 months prior to the 0 month RFA visit (other than cauterization or excision of condyloma(s))
10. Prior ablation or resection therapy consisting of ≥ 75% circumference within the ETZ of anal canal.
11. History of topical therapy (e.g. Imiquimod, 5-FU, Trichloroacetic acid) within the ETZ within 3 months prior to the 0 month RFA visit
12. Hemorrhoids > grade III
13. Fecal incontinence
14. Concurrent disease requiring systemic immunosuppression therapy
15. Concurrent malignancy requiring systemic therapy
16. Life expectancy < 2 years
17. Subject is on a platelet inhibiting agent (i.e. Aspirin, Clopidogrel, NSAIDS) and/or anti-thrombotic agent (Heparin, Warfarin) and unable to discontinue 7 days before and after treatment for 14 days total.

    * Exception: Aspirin 81 mg PO daily does not need to be discontinued

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laser Surgery Care, New York, New York, United States

REFERENCES:
- [Derived] Goldstone RN, Hasan SR, Goldstone SE. Brief Report: Radiofrequency Ablation Therapy for Anal Intraepithelial Neoplasia: Results From a Single-Center Prospective Pilot Study in HIV+ Participants. J Acquir Immune Defic Syndr. 2017 Dec 1;76(4):e93-e97. doi: 10.1097/QAI.0000000000001535. PMID 28857936

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiofrequency Ablation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: subjects who have biopsy-proven HSIL and are HIV-negative or HIV-positive.
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Related Adverse Events
Description: Adverse event : Device relationship - Definite, Probable, Possible
Time Frame: Within 12 months post RFA
Measure: Number; unit: number of participants
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 10
number of participants
  Definite | 1
  Probable | 1

2. Secondary Outcome: Subject Tolerability: Post -Ablation Anal Pain
Description: Median post-ablation anal pain from 10 patients' survey after RFA treatment. Anal pain scale range: 0-10 (minimum pain=0, maximum pain=10)
Time Frame: within 4 weeks post RFA
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 10
units on a scale | 5 [2 to 9]

3. Secondary Outcome: Quality of Life Assessment: Subject Score for Worry About Anal Canal Condition
Description: Median from subject scores for worry about anal canal condition at 0-2 weeks prior to RFA treatment and after 9-12 months post RFA. Median scale range: 0-10 (minimum concern=0, maximum concern=10)
Time Frame: 0-2 weeks Prior RFA and after 9-12 months post RFA
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Radiofrequency Ablation
Number analyzed (Participants) | 10
units on a scale
  0-2 weeks Prior RFA | 4.5 [0 to 8]
  9 to 12 months post RFA | 0.5 [0 to 5]

ADVERSE EVENTS:
Arm/Group | Radiofrequency Ablation
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Ablation (N=10)
Anal Stricture (Injury, poisoning and procedural complications) | 1 (1)
External thrombosed Hemorrhoids (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less